CLINICAL TRIAL: NCT04313426
Title: Evaluating Community-Based Pain Self-Care Using Integrative Yoga Therapy (IYT): Quasi Experimental Study
Brief Title: Chronic Pain Self-Management With Integrative Yoga Therapy (IYT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarogyam UK (Other)
Collaborators: Hindu Swayamsevak Sangh (UK) (Unknown); Leicester Ageing Together (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AU05
Record Dates: First submitted 2020-03-17; First posted 2020-03-18 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Chronic Pain; Chronic Nonmalignant Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrative Yoga Therapy (Experimental): Self managed Yoga based practices were included in one to one sessions for 6-sessions.
  Interventions: Other: Integrative Yoga Therapy

INTERVENTIONS:
Other: Integrative Yoga Therapy — Integrative Yoga Therapy included personalised yoga therapy sessions including their standard care, yoga movements, relaxation, meditation, breathing practices and yoga counselling sessions.

SUMMARY:
The purpose of this study was to evaluate efficacy of chronic pain self-management program in community settings to adopt Integrative Yoga Therapy (IYT).

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old.
* having a chronic pain of more than 3 months of duration, no matter the aetiology.
* Capable of understanding and giving written informed consent.
* Significant levels of distress and disability related to the pain at the beginning of treatment

Exclusion Criteria:

* Intelectual disability or cognitive impairment
* Planning to move out of area
* Serious mental illness
* Drugs or substance abuse in the last 6 months
* Post surgery or scheduled for surgery
* Cancer related pain

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | From baseline to 6-week post intervention
  Analogical Visual Scale from 0 to 10 scores where 0 describes no pain and 10 worst pain.

SECONDARY OUTCOMES:
Anxiety and Depression | From baseline to 6-week post intervention
  Hospital Anxiety and Depression Scale (HADS). 14 item, 7 each of anxiety and depression. Each item score between 0-3.
Satisfaction with the treatment | From Baseline to 6-week post intervention
  Satisfaction with the treatment (CRES-4) 4 questions.
General Quality of Life | From baseline to 6-week post intervention
  Nottingham Health Profile score between 0 to 100 where 0 is best and 100 is worst

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Principal Investigator — Aarogyam UK; Jaydeep Joshi, BAMS, Study Director — Aarogyam UK; Usha Solanki, Study Chair — Hindu Swayamsevak Sangh; Bharti Mistry, Study Chair — Leicester Ageing Together
Locations (1):
- Karyalaya, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided